CLINICAL TRIAL: NCT02059733
Title: Developing a Novel Imaging Biomarker in the Differential Diagnosis of Parkinson's Disease and Parkinsonism by 18F-DTBZ PET
Brief Title: Developing a Novel Imaging Biomarker in the Differential Diagnosis of Parkinson's Disease and Parkinsonism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yi-Hsin Weng, Associate Professor, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 101-1273A
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Parkinson's Disease
Keywords: 18F-DTBZ
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 18F-DTBZ for Parkinson's Disease and parkinsonism (Experimental): This study will compare the brain uptake of 18F- DTBZ in 20 patients with PD, 20 patients with MSA, 20 patients with PSP, 20 patients with CBS, and 20 patients with VaP, 20 patients with ET, and 10 patients with DT.
  Each evaluable subject involved in this study must fulfill all the inclusion and exclusion criteria according the subject grouping, each subject will have 3 visits in this study. Safety measurement will be evaluated by medical history, vital signs, physical examinations, laboratory examinations and collecting of adverse events.
  Interventions: Drug: 18F-DTBZ

INTERVENTIONS:
Drug: 18F-DTBZ — During this study, subjects will receive a single i.v. administration of approximately 10 mCi 18F-DTBZ immediately prior to imaging.
  The proposed dose for this study is based on our phase I study. At the proposed human dose of 10 mCi, the whole body effective dose (ED) will be approximately 680 mrem. The estimated human ED is expected to be comparable to or below the range of other approved brain imaging agents, such as 18F-FDG.

SUMMARY:
This study will compare the brain uptake of 18F- DTBZ in 20 patients with PD, 20 patients with MSA, 20 patients with PSP, 20 patients with CBS, and 20 patients with VaP, 20 patients with ET, and 10 patients with DT.

DETAILED DESCRIPTION:
Study duration is expected to be completed in a period of 4 year. This study is a uncontrolled, open-label, non-randomized, parallel, and cross-sectional study. Total 130 subjects, including 20 patients with PD, 20 patients with MSA, 20 patients with PSP, 20 patients with CBS, 20 patients with VaP, 20 patients with ET, and 10 patients with DT, will be enrolled.

Each evaluable subject involved in this study must fulfill all the inclusion and exclusion criteria according the subject grouping, each subject will have 3 visits in this study, as one screening visit, one imaging visit, and one safety evaluation visit.

Safety measurement will be evaluated by medical history, vital signs, physical examinations, laboratory examinations and collecting of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Twenty subjects with a diagnosis of PD whom must:

   i. Male or female patients, age range 20~80. ii. Patients should be fulfilled "UK Parkinson's Disease Society Brain Bank Criteria for the Diagnosis of PD" (Appendix I).

   iii. Patients who provide a written informed consent prior to study entry. If the patient is incapable of informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm assent).
2. Twenty subjects with a diagnosis of MSA whom must:

   i. Male or female patients, age range 20~80. ii. Patients should be fulfilled the Consensus diagnostic criteria of "possible" or "probable" MSA14 (Appendix I).

   iii. Patients who provide a written informed consent prior to study entry. If the patient is incapable of informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm assent).
3. Twenty subjects with a diagnosis of PSP whom must:

   i. Male or female patients, age range 20~80. ii. Patients should be fulfilled the NINDS-SPSP clinical criteria for the diagnosis of PSP " as possible" or "probable" PSP55 (Appendix III).

   iii. Patients who provide a written informed consent prior to study entry. If the patient is incapable of informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm assent).
4. Twenty subjects with a diagnosis of CBS whom must:

   i. Male or female patients, age range 20~80. ii. Patients should be fulfilled the"Mayo Clinic proposed criteria for the diagnosis for corticobasal syndrome"56 (Appendix I).

   iii. Patients who provide a written informed consent prior to study entry. If the patient is incapable of informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm assent).
5. Twenty subjects with a diagnosis of VaP whom must:

   i. Male or female patients, age range 20~80. ii. Patients should be fulfilled the clinical diagnostic criteria of vascular parkinsonism. (Appendix I).

   iii. Patients who provide a written informed consent prior to study entry. If the patient is incapable of informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm assent).
6. Twenty subjects with a diagnosis of ET whom must:

   i. Male or female patients, age range 20~80. ii. Patients should be fulfilled the "The Consensus Criteria of the MDS on Essential Tremor"30. (Appendix I).

   iii. Patients who provide a written informed consent prior to study entry. If the patient is incapable of informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm assent).
7. Ten subjects with a diagnosis of DT whom must:

   i. Male or female patients, age range 20~80. ii. Patients should be fulfilled the "The Consensus Criteria of the MDS on Dystonic Tremor"30. (Appendix I).

iii. Patients who provide a written informed consent prior to study entry. If the patient is incapable of informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm assent).

Exclusion Criteria:

1. Pregnant or becoming pregnant during the study (as documented by pregnancy testing at screening or at any date during the study according to the PI discretion) or current breast feeding..
2. Any subject who has a clinically significant abnormal laboratory values, and/or clinically significant or unstable medical or psychiatric illness.

   i. Clinically significant hepatic, renal, pulmonary, metabolic, or endocrine disturbances.

   ii. Current clinically significant cardiovascular disease. (cardiac surgery or myocardial infarction within the last 6 months; unstable angina; decompensated congestive heart failure; significant cardiac arrhythmia; congenital heart disease.
3. History of drug or alcohol abuse within the last year, or prior prolonged history of abuse.
4. History or presence of QTc prolongation.
5. History of intracranial operation, including thalamotomy, pallidotomy, and/or deep brain stimulation.
6. Any documented abnormality in the brain by CT or MRI of brain, which might contribute to the motor function, such as hydrocephalus and encephalomalacia, will be excluded. Mild cortical atrophy and non-specific white matter changes will be allowed.
7. Patients who have the evidence of secondary parkinsonism or other neurodegenerative diseases, such as spinocerellar atrophy (SCA), Wilson's disease, hydrocephalus , serious head injury and definite history of neurotoxin exposure, are excluded.
8. History of allergy to radioligands that contain 18F isotope.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-02; Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Analyzing the differences of monoaminergic degeneration between each group by comparing the SUVR of 18F- DTBZ measured by the VOIs methods in each brain region. | 4 years
  During this study, subjects will receive a single i.v. administration of approximately 10 mCi 18F-DTBZ immediately prior to imaging.
  The proposed dose for this study is based on our phase I study. At the proposed human dose of 10 mCi, the whole body effective dose (ED) will be approximately 680 mrem. The estimated human ED is expected to be comparable to or below the range of other approved brain imaging agents, such as 18F-FDG.

SECONDARY OUTCOMES:
Statistical parametrical mapping will be performed to compare the early-phase and delayed-phase imaging of 18F- DTBZ PET in each group. | 4 years
  Statistical parametrical mapping (SPM) will be performed to compare the early-phase (cerebral perfusion) and delayed-phase (monoaminergic system) imaging of 18F- DTBZ PET in each group. The capability of 18F- DTBZ PET imaging as an imaging biomarker in differentiating PD and PM will be also investigated.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memory Hospital, Taoyuan District, Taiwan